CLINICAL TRIAL: NCT00421343
Title: Secondary Prevention of Osteoporosis: A Window of Opportunity in the Acute Rehabilitation Setting
Brief Title: Secondary Prevention of Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Merck Sharp & Dohme LLC (Industry); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Sarah Berry, Research Scientist, Hebrew SeniorLife
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG0074; 5T32AG023480-03 (NIH)
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Results first posted 2011-06-10 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Osteoporosis
Keywords: disease/disorder proneness/risk; osteoporotic fractures; accidental falls; aging
MeSH Terms: conditions — Osteoporosis; Disease Susceptibility; Osteoporotic Fractures | interventions — Alendronate; Cholecalciferol; Fumigant 93; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment for osteoporosis and falls (Other): calcium, vitamin D, a weekly oral bisphosphonate, and falls prevention measures. No comparator group. All participants received the same intervention
  Interventions: Drug: alendronate with cholecalciferol; Drug: calcium carbonate with cholecalciferol; Behavioral: Falls prevention measures

INTERVENTIONS:
Drug: alendronate with cholecalciferol — alendronate 70mg /cholecalciferol 2800IU orally once weekly
  Other Names: Fosamax Plus D®
Drug: calcium carbonate with cholecalciferol — calcium carbonate 500mg /cholecalciferol 200IU orally twice daily
  Other Names: Os-Cal with extra D
Behavioral: Falls prevention measures — personalized exercises, home safety evaluation, referral to an eye doctor if needed, review of medications

SUMMARY:
The purpose of this study is to develop and implement an evidence based protocol for the secondary prevention of osteoporotic fractures and falls, and to determine how compliance with this intervention improves muscle strength and functional status following a fracture.

DETAILED DESCRIPTION:
Following a fracture, few persons are screened or treated for osteoporosis (Feldstein et al). It is not surprising, then, that the risk of future osteoporotic fractures remains high. Although little data exists on the secondary prevention of osteoporosis, calcium, vitamin D, and bisphosphonates have all been shown to be effective in the primary prevention of osteoporotic fractures, and they are likely beneficial in reducing secondary fractures as well. Targeting falls prevention is another approach that is likely effective in reducing the risk of fracture.

In the U.S., acute rehabilitation (rehab) settings offer a unique environment to initiate osteoporotic therapy. Therefore, this study will develop and implement evidence based interventions for the secondary prevention of osteoporotic fractures in the acute rehab setting with the following objectives:

Specific Aim I: Assess overall compliance with pharmacological and non-pharmacological interventions initiated in an acute rehab setting following a fragility fracture. Hypothesis: Non-compliant participants are less likely to show improvement in functional status, muscle strength, or vitamin D levels following the intervention.

Specific Aim II: Describe the incidence of fragility fractures and falls in participants at 6-months and one-year following the osteoporotic intervention introduced during acute rehab. Hypothesis: Similar to community based studies, a number of participants will go on to experience repeat falls and resulting fractures within one-year of follow-up. Compliant participants are less likely to experience falls and fractures.

Specific Aim III: Confirm the high prevalence of vitamin D deficiency in a rehab setting. Describe the relationship between changes in vitamin D levels in participants between baseline and 6-month follow-up and changes in functional outcomes. Hypothesis: There will be a direct association between a change in vitamin D levels and a change in functional status.

Consecutive individuals admitted with the primary or secondary diagnosis of fracture in the rehabilitation unit of Hebrew Rehabilitation Center will be offered enrollment. All participants enrolled will receive the same intervention: calcium, vitamin D, a weekly oral bisphosphonate, and falls prevention interventions. Specific interventions for preventing falls include optimization of visual acuity, a review of medications associated with falls, personalized exercises to improve strength and balance, and a home hazards safety evaluation when indicated.

All participants will have their functional status, muscle strength, and vitamin D level measured at baseline during their rehab stay. At the six-month follow-up, a home visit will be performed for all participants to again assess functional status, muscle strength, vitamin D level, satisfaction with the intervention, and reasons for non-compliance. A history of interim falls and fractures will be collected by telephone interviews, during home nursing visits, and during the exit 6-month visit.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to rehab unit with the primary or secondary diagnosis of fracture
* English speaking
* Cognitively able to provide consent or health care proxy available and willing to provide consent
* Willing to cooperate

Exclusion Criteria:

* Pathologic or periprosthetic fractures
* Creatinine clearance less than 15ml/minute
* Severe hypocalcemia
* Esophageal stricture or achalasia
* Taking other treatment for osteoporosis besides calcium or vitamin D in the past 6-months
* History of kidney stones in the past 6-months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah D Berry, MD, MPH, Principal Investigator — Harvard University, Hebrew Rehabilitation Center
Locations (1):
- Hebrew SeniorLife, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kamel HK. Secondary prevention of hip fractures among the hospitalized elderly: are we doing enough? J Clin Rheumatol. 2005 Apr;11(2):68-71. doi: 10.1097/01.rhu.0000158545.26370.5c. PMID 16357705
- [Background] Dawson-Hughes B, Harris SS, Krall EA, Dallal GE. Effect of calcium and vitamin D supplementation on bone density in men and women 65 years of age or older. N Engl J Med. 1997 Sep 4;337(10):670-6. doi: 10.1056/NEJM199709043371003. PMID 9278463
- [Background] Cummings SR, Black DM, Thompson DE, Applegate WB, Barrett-Connor E, Musliner TA, Palermo L, Prineas R, Rubin SM, Scott JC, Vogt T, Wallace R, Yates AJ, LaCroix AZ. Effect of alendronate on risk of fracture in women with low bone density but without vertebral fractures: results from the Fracture Intervention Trial. JAMA. 1998 Dec 23-30;280(24):2077-82. doi: 10.1001/jama.280.24.2077. PMID 9875874
- [Background] Gillespie LD, Gillespie WJ, Robertson MC, Lamb SE, Cumming RG, Rowe BH. Interventions for preventing falls in elderly people. Cochrane Database Syst Rev. 2003;(4):CD000340. doi: 10.1002/14651858.CD000340. PMID 14583918
- [Background] Feldstein A, Elmer PJ, Orwoll E, Herson M, Hillier T. Bone mineral density measurement and treatment for osteoporosis in older individuals with fractures: a gap in evidence-based practice guideline implementation. Arch Intern Med. 2003 Oct 13;163(18):2165-72. doi: 10.1001/archinte.163.18.2165. PMID 14557214

RESULTS

PARTICIPANT FLOW:
Groups:
- Osteoporosis Medication: Everyone received 1000 mg calcium per day plus vitamin D and alendronate 70mg per week.
Period: Overall Study
Arm/Group | Osteoporosis Medication
Started | 29
Completed | 23
Not Completed | 6
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Osteoporosis Medication
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 80 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Number Adherent With the Intervention
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Osteoporosis Medication
Number analyzed (Participants) | 29
participants | 29

2. Secondary Outcome: Reasons for Non-willingness to Particiapte and Non-adherence With Intervention
Description: We asked participants who would not participate the primary reason for non-particiaption. We also asked participants who were not adherent with recommendations what the primary reason ws for non-adherence.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Osteoporosis Medication
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osteoporosis Medication (N=29)
death (Injury, poisoning and procedural complications) | 1 (1) — One subject experienced a fall resulting in a high cervical injury and death, not related to study intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No